CLINICAL TRIAL: NCT01873430
Title: The Sun Protective Effect of Melatonin: a Randomized, Placebo-controlled, Double-blind Study on Healthy Volunteers
Brief Title: The Sun Protective Effect of Melatonin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Cecilie Scheuer, Research scholar, medical student, Herlev Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: 2013-000629-30
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Sunburn
Keywords: Melatonin; Sunburn; Erythema; Sunlight; Ultraviolet rays
MeSH Terms: conditions — Sunburn; Erythema | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Melatonin: Melatonin cream 2,5% (Active Comparator): One square on the back of each volunteers will be randomized to have the above mentioned dose of melatonin cream applied
  Interventions: Drug: Melatonin
- Melatonin: Melatonin cream 0,5% (Active Comparator): One square on the back of each volunteers will be randomized to have the above mentioned dose of melatonin cream applied.
  Interventions: Drug: Melatonin
- Melatonin: Melatonin cream 12,5% (Active Comparator): One square on the back of each volunteers will be randomized to have the above mentioned dose of melatonin cream applied.
  Interventions: Drug: Melatonin
- placebo cream (Placebo Comparator): One square on the back of each volunteers will be randomized to have placebo cream (vehicle) applied.
- No treatment (No Intervention): One square on the back of each volunteers will be randomized to receive no treatment.

INTERVENTIONS:
Drug: Melatonin
  Arms: Melatonin: Melatonin cream 0,5%; Melatonin: Melatonin cream 12,5%; Melatonin: Melatonin cream 2,5%

SUMMARY:
The aim of this study is to investigate the sun protective effect of melatonin, when used as a cream applied before sun exposure.

Sun exposure induces erythema as indication of an inflammatory reaction in the skin. It is proven that the amount of free radicals in the skin are increased by UV exposure. Furthermore, it is known that melatonin is a potent antioxidant. It is hypothesized that melatonin can be protective against the UV induced release of free radicals by acting as a radical scavenger and thereby protect against UV-induced cellular damage.

DETAILED DESCRIPTION:
This study investigates the sun protective effect of melatonin when used as a creme applied before sun exposure.

The study is a randomized, placebo-controlled, double-blinded study conducted on healthy volunteers. The volunteers will have 5 squares of 8 cm*8 cm on their backs, which each will be randomized to receive one of following: melatonin cream 0,5%; melatonin cream 2,5%; melatonin cream 12,5%; placebo cream (vehicle) and no treatment.

After randomization and received treatment the volunteers will be exposed to strong midday sun (UV-index of approximately 9) for 40 minutes.

The outcomes parameters (degree of erythema and pain sensation) are measured at baseline and 1,4,8 and 24 hours post exposure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers of both sexes.
* Skin type 1-3 according to Fitzpatrick skin type scale.
* No sun exposure on skin area tested in the study 4 weeks prior to the study.

Exclusion Criteria:

* Active skin disease
* Participant that do not react to the given sun exposure with a change in a-value >5 are excluded from the data.
* Pregnancy
* Previous malignant or pre malignant skin disease.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-05; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Reduction of erythema assessed by digital image analysis (Image J) after treatment with melatonin/placebo before sun exposure. | Primary outcome is assessed at: baseline and 1,4,8 and 24 hours post exposure
  The alpha value measured in a "color space converted" image will represent the degree of erythema

SECONDARY OUTCOMES:
Testing for primary hyperalgesia in the sun exposed area with Pin-Prick monofilaments. Testing for primary hyperalgesia in the sun-exposed area with Pin-Prick monofilaments. | The secondary outcome is assessed at: baseline and 1,4,8 and 24 hours post exposure.

OTHER OUTCOMES:
Visual inspection of erythema using Frosch-Klingman scale. | This secondary outcome is assessed at: baseline and 1,4,8 and 24 hours post exposure

CONTACTS AND LOCATIONS:
Overall Officials: Cecilie Scheuer, Research Scholar, Principal Investigator — Gastroenheden, Herlev Hospital
Locations (1):
- Gastroenheden, Herlev Hospital, Herlev, Herlev, Denmark